CLINICAL TRIAL: NCT03019224
Title: Effects of Desensitizing Dentifrices on the Reduction of Pain Sensitivity Caused by In-office Dental Whitening: Double Blind Controlled Clinical Study
Brief Title: Effects of Desensitizing Dentifrices on the Reduction of Pain Sensitivity Caused by In-office Dental Whitening
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Josué Junior Araujo Pierote, Principal Investigator, University of Campinas, Brazil
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 104/2015
Record Dates: First submitted 2016-12-19; First posted 2017-01-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Tooth Whitening; Sensitivity
Keywords: Tooth whitening; Dentifrice; Sensitivity
MeSH Terms: conditions — Hypersensitivity | interventions — Hydrogen Peroxide

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Placebo Comparator): The use of desensitizing dentifrice [Sucralose (S) Control dentifrice)] in plastic tray.
  Interventions: Procedure: Selection and preparation of the volunteers; Procedure: Evaluation of the tooth color; Procedure: Relative isolation; Procedure: Gingival protection barrier; Procedure: Application of desensitizing gel; Drug: Hydrogen peroxide; Procedure: Used a dentifrice
- Group 2 (Experimental): The use of desensitizing dentifrice [Sodium fluoride (FS) with 1450ppm of fluorine (Close up triple, Unilever)] in plastic tray.
  Interventions: Procedure: Selection and preparation of the volunteers; Procedure: Evaluation of the tooth color; Procedure: Relative isolation; Procedure: Gingival protection barrier; Procedure: Application of desensitizing gel; Drug: Hydrogen peroxide; Procedure: Used a dentifrice
- Group 3 (Experimental): The use of desensitizing dentifrice [Arginine, calcium carbonate (ACC) and sodium monofluorophosphate with 1450 ppm fluorine (Colgate sensitive pro-relief, Colgate-Palmolive)] in plastic tray.
  Interventions: Procedure: Selection and preparation of the volunteers; Procedure: Evaluation of the tooth color; Procedure: Relative isolation; Procedure: Gingival protection barrier; Procedure: Application of desensitizing gel; Drug: Hydrogen peroxide; Procedure: Used a dentifrice
- Group 4 (Experimental): The use of desensitizing dentifrice [Sodium fluoride based dentifrice with 1450 ppm of fluorine associated with 5% potassium nitrate] in plastic tray.
  Interventions: Procedure: Selection and preparation of the volunteers; Procedure: Evaluation of the tooth color; Procedure: Relative isolation; Procedure: Gingival protection barrier; Procedure: Application of desensitizing gel; Drug: Hydrogen peroxide; Procedure: Used a dentifrice

INTERVENTIONS:
Procedure: Selection and preparation of the volunteers — Patients who sought the postgraduate dental clinic for whitening were invited to participate in the study. They were informed by the researcher (dentist) about all the aspects of the study and who might participate or discontinue the participation at any moment during the treatment. In addition, it was clarified that their participation was voluntary and refusal to participate would not result in any penalty or loss of benefits.
Procedure: Evaluation of the tooth color — The evaluation of the tooth color was performed by using a spectrophotometer (Easyshade, Vident, Brea, CA, USA). The color was analysed with the tooth hydrated before of the start the first whitening session and one week after.
  The spectrophotometer was always used in the same position by a silicon guide, which was prepared with dental arch molds by adding high viscosity vinyl polysiloxane material (Express XT, 3M ESPE, Sumaré, SP, Brazil). After polymerization, an opening was made in the mold corresponding to the buccal surface of the upper central incisors, allowing the color of the tooth to be evaluated with the tip of the spectrophotometer at the height of the middle third.
Procedure: Relative isolation — The clinical procedures were performed under relative isolation using lip retractor (Arcflex, FGM, Joinville, SC, Brazil) and dental cotton rollers to apply a gingival protection barrier (Top Dam, FGM, Joinville, SC, Brazil) extending from right first molar to left first molar in both arches.
Procedure: Gingival protection barrier — The gingival protection barrier was placed over the margins and gingival papilla corresponding to the areas receiving the whitening gel with approximately 3 mm in height and photopolymerized for 20 seconds in each group of three tooth. Photo-activation was performed with high power LEDs (light intensity = 600mw / cm²) (RadiiCal, São Paulo, SP, Brazil).
Procedure: Application of desensitizing gel — The desensitizing gel containing 5% potassium nitrate associated with 2% sodium fluoride (Desensibilize KF 2%, FGM, Joinville, SC, Brazil) was applied with a microbrush (Brush KG, KG Sorensen, Cotia, SP) on the buccal surface from right first molar to left first molar in both arches and remaining for 10 minutes. Then, the desensitizer was then removed with water jet and disposable plastic suction cannula.
Drug: Hydrogen peroxide — The handling of 35% hydrogen peroxide (Whiteness HP, FGM, Joinville, SC, Brazil) followed the manufacturer's recommendations, which consisted of mixing 3 drops of 35%hydrogen peroxide for 1 drop of thickener, with this mixture being sufficient for application to at least three tooth. The gel remained in contact with the buccal surface of the tooth for 15 minutes and was removed with disposable plastic suction cannula and water wash. This procedure was performed three times per clinical session. The volunteers underwent three whitening clinical sessions with one week interval between them.
Procedure: Used a dentifrice — Among the clinical whitening sessions, each volunteer used an unidentified dentifrice corresponding to their experimental group, which was previously defined by means of a draw made by a dentist who did not participate in the study. Thus, the researcher (dentist) who provided the dentifrice and the volunteer were not aware of which experimental group belonged (i.e. double blind).

SUMMARY:
Introduction: The pain sensitivity associated with whitening is the main problem reported by patients during dental whitening, and the use of desensitizing dentifrices is an alternative for the treatment of sensitivity.

Objective: To evaluate clinically the influence of desensitizing dentifrices applied through a plastic tray, reducing the pain sensitivity and color variation caused by the technique of in-office dental whitening, through a controlled double-blind clinical study.

Methods: A longitudinal prospective study was conducted with 48 individuals, 18 years and 30 years of age, without gender distinction, who underwent in-office dental whitening using 35% hydrogen peroxide (Whiteness HP, FGM, Joinville , SC, Brazil) in three clinical sessions with a one-week interval between them. The volunteers used in the night for each bleaching session a plastic tray for 4 hours containing one of the dentifrices related to the experimental groups: Group 1 (Control) - Sucralose (S) (Biotype - Manipulation pharmacy); Group 2 (Active control) - Sodium fluoride (FS) with 1450ppm of fluorine (Close up triple, Unilever); Group 3 - Arginine, calcium carbonate (ACC) and sodium monofluorophosphate with 1450 ppm fluorine (Colgate sensitive pro-relief, Colgate-Palmolive); Group 4 - 5% potassium nitrate (NP) and sodium fluoride with 1450 ppm fluorine (Sensodyne pro-enamel, GlaxoSmithKline). The evaluation of the sensitivity associated with the times of use of the plastic tray in the first session (S1: sensitivity before the tray, S2: sensitivity after the tray), in the second session (S3: sensitivity before the tray, S4: in the third session (S5: sensitivity before the tray, S6: sensitivity after the tray) used the analog numerical scale with scores from 0 to 10 and for the color evaluation the spectrophotometer (Easyshade, Vident, Brea, CA, Obtaining the data that were used in the CIELab system. The data were submitted to the multivariate analysis of variance (MANOVA) with repeated measurements and Lambda Wilks test with a 5% probability level to differentiate the groups. In addition, the factorial variance analysis (ANOVA) in one criterion was applied. Values of p <0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* age of 18 years or older
* good oral and general health
* hygid anterior tooth with color shade higher than A2 on the Vita Classic scale (VITA Zahnfabrink, Bad Säckingen, Germany).

Exclusion Criteria:

* smoking, pregnancy or breastfeeding
* previous dental whitening
* para-functional habits
* dentin sensitivity
* anterior tooth with restorations and carious lesions
* non-vital discoloration
* unsatisfactory restorations

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2016-01; Primary Completion 2016-04 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The analysis of the reduction of sensitivity using the toothpaste during whitening. | Through study completion up to 4 weeks placement of the tray.
  For sensitivity analysis was used the numerical analogue scale with scores ranging from 0 to 10.
The evaluation of the tooth color using the toothpaste during whitening. | Through study completion up to 4 weeks placement of the tray.
  For evaluation of the tooth color was performed by using a spectrophotometer. (Easyshade, Vident, Brea, CA, USA). The color was determined by EasyShade device.

IPD SHARING:
Plan to Share IPD: Undecided